CLINICAL TRIAL: NCT01865721
Title: Optimizing the Use of Entonox® During Screening Colonoscopy: an Open Randomised Controlled Trial
Brief Title: Optimizing the Use of Entonox® During Screening Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH16359; 2012-003342-33 (EudraCT Number)
Record Dates: First submitted 2013-05-21; First posted 2013-05-31 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Bowel Cancer Screening; Analgesia; Entonox; Colonoscopy
Keywords: Bowel cancer screening; Analgesia; Entonox; Pain; Side effects; Colonoscopy
MeSH Terms: conditions — Agnosia; Pain | interventions — Entonox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous administration of Entonox (Active Comparator): Patients randomized to this arm will be asked to inhale Entonox throughout the insertion phase of colonoscopy
  Interventions: Drug: Entonox
- As required administration of Entonox (Active Comparator): Patients randomised to this arm will be asked to use Entonox if and when they have pain
  Interventions: Drug: Entonox

INTERVENTIONS:
Drug: Entonox — Entonox will be used according to the allocated method

SUMMARY:
This study will randomise patients undergoing screening colonoscopy to receive Entonox either continuously or as required.

Both these methods are used in the published studies of Entonox and in clinical practice.

Null hypothesis There will be no difference in pain levels between these two methods of Entonox administration

ELIGIBILITY:
Inclusion Criteria:

* Having a bowel cancer screening programme colonoscopy

Exclusion Criteria:

* Contraindications to Entonox
* Previous bowel resections

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pain scores | Day 1: Prior to discharge from endoscopy department
  Patients will be asked about their overall recollection of pain on a 10 point numerical ratings scale prior to discharge

SECONDARY OUTCOMES:
Pain scores | Day 1-4: Prior to discharge and 1-3 days later
  Patients will be asked about their experience of pain during colonoscopy. In addition patients will be asked about their overall recollection of pain immediately after colonoscopy and 1-3 days following colonoscopy.
Use of analgesia and sedation | Day 1: During colonoscopy
  Patients additional use of sedation and analgesia will be compared in each treatment arm
Patients satisfaction | Day 1-4: Prior to discharge and 1-3 days later
  Patients will be asked about their overall level of satisfaction immediately prior to discharge and 1-3 days later
Willingness to have a repeat colonoscopy | Day 1: Prior to discharge
  Patients will be asked about their willingness to have a repeat colonoscopy prior to discharge and 1-3 days following colonoscopy
Side Effects | Day 1: During colonoscopy
  Patients will be asked about the presence of side effects during colonoscopy. This will be quantified according to whether it limited the use Of Entonox.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Riley, MB ChB, Principal Investigator — Sheffield Teaching Hospital
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Ball AJ, Din S, Donnelly M, Riley SA. A randomized controlled trial comparing continuous and as-required nitrous oxide use during screening colonoscopy. Eur J Gastroenterol Hepatol. 2015 Mar;27(3):271-8. doi: 10.1097/MEG.0000000000000281. PMID 25629571